CLINICAL TRIAL: NCT03193957
Title: An Open-label, Single-arm, Multicentre Clinical Study to Evaluate the Usability and Safety of the Autoinjector and Pre-filled Syringe of SB4 in Subjects With Rheumatoid Arthritis
Brief Title: An Multicentre Clinical Study to Evaluate the Usability and Safety of the Autoinjector and Pre-filled Syringe of SB4 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SB4-G21-RA
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB4 (Experimental): SB4 (etanercept) 50 mg/mL
  Interventions: Drug: Etanercept; Device: Autoinjector

INTERVENTIONS:
Drug: Etanercept — Etanercept PFS and Autoinjector
Device: Autoinjector — Autoinjector

SUMMARY:
A study comparing the usability of the Autoinjector and Pre-filled Syringe of SB4 in Subjects with Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are male or female aged 18-55 years at the time of signing the informed consent form.

Exclusion Criteria:

* Have been treated previously with monoclonal antibody agent including any tumour necrosis factor inhibitor except SB4.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-08-03 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
The change in Injection site pain score at immediately post injection (within 1 minute) | at Week 1 and Week 3
  The change in injection site pain score at immediately post injection (within 1 minute) using an 11-point visual numeric scale

CONTACTS AND LOCATIONS:
Locations (1):
- AI Centrum Medyczne, Poznan, Poland

REFERENCES:
- [Derived] Rho YH, Rychlewska-Hanczewska A, Sliwowska B, Kim TH. Usability of Prefilled Syringe and Autoinjector for SB4 (An Etanercept Biosimilar) in Patients with Rheumatoid Arthritis. Adv Ther. 2019 Sep;36(9):2287-2295. doi: 10.1007/s12325-019-01027-z. Epub 2019 Aug 1. PMID 31372961